CLINICAL TRIAL: NCT03908229
Title: Trainee Participation Increases Colon Adenoma Detection Rate: a Randomized Controlled Trial
Brief Title: Trainee Participation Increases Colon Adenoma Detection Rate
Acronym: ADR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti di Foggia (Other)
Responsible Party: Principal Investigator, Antonio Facciorusso, Assistant Professor of Gastroenterology, Ospedali Riuniti di Foggia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ADR01
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trainee colonoscopy (Experimental): In the investigation arm colonoscopy will be performed by gastroenterology fellows. The fellows will always start the case and proceed generally until they are unable to make further progress despite "coaching" from the staff attending.
  During the procedures with fellows, the staff attending will always actively participate in the entire procedure and assess for the presence of any lesions.
  Interventions: Procedure: Trainee colonoscopy
- Experienced physician colonoscopy (Active Comparator): In the control arm all colonoscopy will be performed by full-time board-certified gastroenterologists who have each done more than 5000 colonoscopy examinations.
  Interventions: Procedure: Experienced physician colonoscopy

INTERVENTIONS:
Procedure: Trainee colonoscopy — Colonoscopy performed by trainee
  Arms: Trainee colonoscopy
Procedure: Experienced physician colonoscopy — Experienced physician colonoscopy
  Arms: Experienced physician colonoscopy

SUMMARY:
Previous studies that examined whether the presence of an additional observer, more specifically a GI fellow, during colonoscopy can enhance detection of all polyps and adenomas yielded conflicting results. Of note, all of the aforementioned studies were retrospective and robust evidence derived from well-designed randomized controlled trials are lacking.

The study objective is to examine whether fellow participation during screening, surveillance, or diagnostic colonoscopy influence overall, size-specific, or location-specific adenoma or polyp detection rate.

It will be planned to enroll 812 patients (406 per arms) within 1 year. Adenoma detection rate will be the primary outcome.

DETAILED DESCRIPTION:
Background Colonoscopy is instrumental in colon cancer prevention as through polypectomy it may interfere with the adenoma-carcinoma sequence, thus resulting in a clear survival benefit.

However, not all adenomatous polyps are identified during a colonoscopy. The overall false-negative ("miss") rate for colonic adenomas is estimated to be as high as 24%, according to studies of same-day, tandem colonoscopies. In addition, flat and depressed lesions often remain undetected during white-light colonoscopy.

Low-cost optimization of existing resources, such as use of a second observer or water-aided colonoscopy, were recently found to be able to significantly increase colon adenoma detection rate (ADR).

Previous studies that examined whether the presence of an additional observer, more specifically a GI fellow, during colonoscopy can enhance detection of all polyps and adenomas yielded conflicting results. Of note, all of the aforementioned studies were retrospective and robust evidence derived from well-designed randomized controlled trials (RCTs) are lacking.

.

Technical procedure In the control arm all colonoscopy will be performed by full-time board-certified gastroenterologists who have each done more than 5000 colonoscopy examinations.

In the investigation arm colonoscopy will be performed by gastroenterology fellows. The fellows will always start the case and proceed generally until they are unable to make further progress despite "coaching" from the staff attending.

During the procedures with fellows, the staff attending will always actively participate in the entire procedure and assess for the presence of any lesions.

Colonoscopies will be performed by using only high-definition white-light (HDWL) scopes (Olympus 180 series CF H180).

Bowel preparation will be uniform and consist of 4 L of polyethylene glycol. All detected lesions will be endoscopically removed and samples will be sent to pathologists for histological diagnosis.

Treatment strategy Patients complying with the eligibility criteria will be randomized in a 1:1 fashion to undergo colonoscopy performed by a trainee (under attending physician supervision) or colonoscopy performed by an experienced physician.

Sample size calculation and statistical considerations On the basis of previous retrospective comparative reports, the study is designed to detect an increase in ADR by 8%. Therefore, 812 patients (406 per arm) will be required to have a 80% power to detect the target difference at a 0.05 significance level (two sided). The primary endpoint will be ADR. In order to collect the estimated sample size, up to 1 year of recruiting will be needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing colonoscopy.

Exclusion Criteria:

* Age under 18 years
* Familial history of polyposis syndrome (familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer, juvenile polyposis).
* Incomplete colonoscopy
* Inflammatory bowel disease
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 12 months

SECONDARY OUTCOMES:
Advanced adenoma detection rate | 12 months
Polyp detection rate | 12 months
Sessile serrated adenoma detection rate | 12 months
Adenoma per colonoscopy rate | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale di San Severo, San Severo, Out of USA Or Canada
  - Ospedale di Taranto, Taranto, Out of USA Or Canada
  - Ospedale di Brindisi, Brindisi
  - Ospedali Riuniti Foggia, Foggia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rex DK, Chadalawada V, Helper DJ. Wide angle colonoscopy with a prototype instrument: impact on miss rates and efficiency as determined by back-to-back colonoscopies. Am J Gastroenterol. 2003 Sep;98(9):2000-5. doi: 10.1111/j.1572-0241.2003.07662.x. PMID 14499778
- [Background] Rex DK. Maximizing detection of adenomas and cancers during colonoscopy. Am J Gastroenterol. 2006 Dec;101(12):2866-77. doi: 10.1111/j.1572-0241.2006.00905.x. PMID 17227527
- [Background] Facciorusso A, Triantafyllou K, Murad MH, Prokop LJ, Tziatzios G, Muscatiello N, Singh S. Compared Abilities of Endoscopic Techniques to Increase Colon Adenoma Detection Rates: A Network Meta-analysis. Clin Gastroenterol Hepatol. 2019 Nov;17(12):2439-2454.e25. doi: 10.1016/j.cgh.2018.11.058. Epub 2018 Dec 6. PMID 30529731
- [Background] Gianotti RJ, Oza SS, Tapper EB, Kothari D, Sheth SG. A Longitudinal Study of Adenoma Detection Rate in Gastroenterology Fellowship Training. Dig Dis Sci. 2016 Oct;61(10):2831-2837. doi: 10.1007/s10620-016-4228-9. Epub 2016 Jul 12. PMID 27405989
- [Background] Nishizawa T, Suzuki H, Takahashi M, Kaneko H, Fujiyama Y, Komatsu H, Nagumo H, Tanaka S, Hibi T. Trainee participation during colonoscopy adversely affects polyp and adenoma detection rates. Digestion. 2011;84(3):245-6. doi: 10.1159/000330736. Epub 2011 Sep 7. No abstract available. PMID 21912131
- [Background] Buchner AM, Shahid MW, Heckman MG, Diehl NN, McNeil RB, Cleveland P, Gill KR, Schore A, Ghabril M, Raimondo M, Gross SA, Wallace MB. Trainee participation is associated with increased small adenoma detection. Gastrointest Endosc. 2011 Jun;73(6):1223-31. doi: 10.1016/j.gie.2011.01.060. Epub 2011 Apr 8. PMID 21481861
- [Derived] Facciorusso A, Buccino VR, Tonti P, Licinio R, Del Prete V, Neve V, Di Maso M, Muscatiello N. Impact of fellow participation on colon adenoma detection rates: a multicenter randomized trial. Gastrointest Endosc. 2020 Dec;92(6):1228-1235. doi: 10.1016/j.gie.2020.05.015. Epub 2020 May 17. PMID 32433915